CLINICAL TRIAL: NCT05441319
Title: Investigation of the Effect of Chronic Ankle Instability on Core Stabilization, Dynamic Balance and Agility in Basketball Players of an University
Brief Title: Effect of Chronic Ankle Instability on Core Stabilization, Dynamic Balance and Agility
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Eda Urhun, Master of Science Student, Yeditepe University
Other Study IDs: yeditepe12
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Ankle Sprains; Ankle Injuries; Chronic Ankle Instability
Keywords: chronic ankle instability; ankle instability; core stability; agility; dynamic balance; balance
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic ankle instability group: After completing the evaluation form containing the demographic and clinical characteristics of all participants at their first visit, the Cumberland Ankle Instability Questionnaire (CAIT) scale will be completed and athletes with a CAIT score ≤ 25 will be assigned to the Chronic Ankle Instability Group;
- Control group: Athletes with a score > 25 in the Cumberland Ankle Instability Questionnaire (CAIT) will be included in the Control Group.

SUMMARY:
Ankle sprains are the most common injury in basketball, especially involving repetitive maneuvers such as acceleration, deceleration, jumping, and landing. The incidence of ankle sprain is 40% in female basketball players and 75% in male basketball players. It is also known that chronic ankle instability (CAI) develops in 20-40% of cases. The effects of chronic ankle instability on core stabilization, dynamic balance and agility in basketball players have been investigated in the literature, and it has been stated that more studies are needed on the subject.

The aim of this study is to examine the effects of chronic ankle instability on core stabilization, dynamic balance and agility in basketball players playing in the university team.

The hypothesis of the study is that there is a difference between core stabilization, dynamic balance and agility values of basketball players playing in the university team with and without chronic ankle instability.

DETAILED DESCRIPTION:
Approximately 10% to 28% of all sports injuries are ankle sprains. Ankle sprains are the most common injury in basketball, especially involving repetitive maneuvers such as acceleration, deceleration, jumping, and landing. The incidence of ankle sprain is 40% in female basketball players and 75% in male basketball players. It is also known that chronic ankle instability (CAI) develops in 20-40% of cases. People with CAI have several types of deficits, including decreased ankle range of motion, decreased ankle arthrokinematic quality of movement, problems with postural control and strength, impaired proprioception and neuromuscular control, and altered gait patterns. These problems can cause loss of matches, increase in health expenditures and future injuries in athletes. Postural control disorders that play a role in the regulation of balance have been shown to be common in people with CAI and after acute lateral ankle sprain. Postural control requires somatosensory, visual and vestibular stimuli and appropriate motor response to generate the appropriate balance response. In individuals with CAI, the ankle joint and postural control mechanisms that cannot receive appropriate afferent stimulation and cannot reveal the correct efferent stimulation from the central nervous system are impaired.

Agility, the ability to make rapid changes in the direction of movement, is widely regarded as an important criterion for success in basketball. Agility tests require rapid deceleration, change of direction, and reacceleration during movements. Such activities put athletes in a condition that can force the ankle complex into excessive inversion and plantar flexion, which often causes ankle sprain.

The relationship between chronic ankle instability and athletic performance parameters has been investigated in previous studies. However, the relationship between chronic ankle instability and athletic performance parameters has not yet been fully explained, and it has been stated that more studies are needed on the subject.

Core stability is the motor control and muscle capacity of the lumbopelvic complex. Studies have shown that weakness in the core musculature can predispose an athlete to injury, including ankle sprains. Subjects with a history of lower extremity injuries require more trunk muscle contractions to stabilize the body during dynamic tasks compared to healthy subjects. Therefore, core muscles are an important element to be evaluated in athletes with chronic ankle instability. Although the relationship between chronic ankle instability and the strength of the core muscles has been examined in the literature, the relationship between them has not been fully explained.

In this study, the relationship between chronic ankle instability and core stabilization, dynamic balance and agility in Yeditepe University basketball players will be discussed and the results will be presented.

The power analysis of the research was made using the G*Power 3.1 program. The power of the study was determined as 80%. In a similar study, the mean of the Y balance test in individuals with chronic ankle instability was reported as 86.61, standard deviation of 3.98, and standard deviation of 9.51 in individuals without chronic ankle instability. Based on these values, power analysis was made with the G*Power 3.1 program. As a result of the analysis made with 80% power, the number of participants in the experimental and control groups was determined as 10 for each group.

SPSS (version 22.0) will be used in the data analysis of our research. Quantitative data to be obtained from the research will be shown as mean and standard deviation. Kolmogorov-Smirnov test will be used to test numerical variables for normality. According to the conformity of the obtained data to the normal distribution; If the data is normally distributed (parametric), Independent Sample t-test will be used to compare the two groups. If the data are not normally distributed, the Mann-Whitney U test will be used to compare the two groups. Qualitative data of the groups will be displayed with frequency and percentage values. The statistical significance level will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

1. To be a voluntary participant in the research.
2. To be between the ages of 18-25.
3. Experiencing recurrent sprains with inflammatory symptoms (pain, swelling) for individuals in the study group whose initial history of sprains was at least 1 year prior to the study.
4. Playing in the basketball team for at least 1 season.
5. Having a "feeling of insecurity" and instability in the injured ankle as verified by the Cumberland Ankle Instability Tool (CAIT) score of ≤25 for individuals in the research group.
6. For the individuals in the research group, not having experienced an ankle sprain in the last 1 month.

Exclusion Criteria:

1. History of surgery for musculoskeletal structures in both lower extremities
2. History of fracture in both lower extremities
3. Acute injury of the musculoskeletal structures of other joints of the lower extremity affecting joint function and integrity in the last 3 months
4. Presence of bilateral ankle instability
5. Balance or vestibular disorder
6. Abdominal surgery history
7. To have had a musculoskeletal injury of the waist, back and neck in the last 3 months.
8. To have experienced an ankle injury in the last 1 month.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: It is planned to include athletes aged 18-25, who play in university basketball teams, with and without chronic ankle instability in our study.
  It will include students between the ages of 18-25 who study at Yeditepe University and play in Yeditepe University basketball teams.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Core stabilization- McGill Trunk Muscle Endurance Test. | 8 weeks
  It will be measured with the McGill Trunk Muscle Endurance Test. The McGill Trunk Muscle Endurance Test consists of 4 different positions: trunk anterior flexor test, right and left lateral plank, and trunk posterior extensor test. Before starting the test, participants are given a practice test in which they try to position the correct position for a few seconds, and a practice test in which they try to stay maximally static in each position. The investigator visually determines the end of all tests to ensure test reliability. This researcher uses the "start" and "stop" commands to start and end the test, while the co-investigator records times using a stopwatch.
Dynamic balance- Y Balance Test | 8 weeks
  It will be measured with the Y Balance Test. The test apparatus is placed by measuring 90 degrees and 135 degrees in 3 directions, anterior, posteromedial and posterolateral.Before starting the test, subjects will be allowed to try each aspect 3 times.
  Participants are asked to reach as far as they can without losing their balance. Distances will then be noted. The test is repeated 3 times in each direction. Participants will be given a 15-second rest period after each direction attempt. The average of the 3 repetitions reached for each of the three directions will be recorded. Normalized reach distances for all directions will be calculated by dividing the mean of the 3 measured replicates by the measured lower extremity length extending from the participants' SIAS to the distal apex of the medial malleolus and multiplying by 100.
Agility- T Test | 8 weeks
  It will be measured with the T Test. The T-test consists of 4 contact points formed in a T-shape in an area 10 m long and 10 m wide. It is aimed to complete a series that requires the person to move in different directions and in different ways between these contact points as soon as possible. After three applications, the best test result is recorded in seconds.

SECONDARY OUTCOMES:
Physical functions of athletes with chronic ankle instability | 8 weeks
  It will be assessed with the The Foot and Ankle Ability Measure (FAAM). The Foot and Ankle Ability Measure will be used to measure the physical functions of athletes with chronic ankle instability. The FAAM consists of 29 items that present two separate subscales: "Activity of Daily Living" consisting of 21 questions and "Sports" consisting of 8 questions. Each question is rated from 0 to 4 with 0 "I can't" and 4 "no difficulty". Each subscale has a maximum potential score (84 ADL and 32 Sports subscales). The score for each subscale is divided by the maximum potential score for the subscale and multiplied by 100 to get a percentage. Therefore, the Foot and Ankle Usability Criterion has two subscales (ADL and Sport) with values ranging from 0 to 100, where higher values mean more physical function.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)